CLINICAL TRIAL: NCT04717076
Title: PrevA Study - Evaluation of an App-based Nutritional Concept to Lower Cardiovascular Risk Factors (Focus: Weight Reduction)
Brief Title: PrevA Study - Evaluation of an App-based Nutritional Concept
Acronym: PrevA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Christine Dawczynski,PhD, PhD, Head of Junior Research Group Nutritional Concepts, University of Jena, University of Jena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H11_21
Record Dates: First submitted 2021-01-12; First posted 2021-01-20 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2021-01

CONDITIONS: Reduction of Cardiovascular Risk Factors
Keywords: personalized nutritional concept, weight reduction, mHealth
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- App-based nutritional concept and fitness tracking (Active Comparator): App-based nutritional concept and fitness tracking
  Interventions: Behavioral: App-based nutritional concept and fitness tracking
- Nutritional concept with individual nutritional counselling (Experimental): Nutritional concept with individual nutritional counselling
  Interventions: Behavioral: Nutritional concept with individual nutritional counselling
- Nutritional concept without individual nutritional counselling (Experimental): Nutritional concept without individual nutritional counselling
  Interventions: Behavioral: Nutritional concept without individual nutritional counselling
- Control group (No Intervention): Control group - no intervention

INTERVENTIONS:
Behavioral: App-based nutritional concept and fitness tracking — The App-based nutritional concept based on menu plan, which are personalized according to participants age, gender, physical activity. The App is coupled with a Smartwatch to encourage and track physical activity over the study period.
  Arms: App-based nutritional concept and fitness tracking
Behavioral: Nutritional concept with individual nutritional counselling — Nutritional concept based on personalized menu plans and individual nutritional counselling every four weeks (4 times during the study)
  Arms: Nutritional concept with individual nutritional counselling
Behavioral: Nutritional concept without individual nutritional counselling — Nutritional concept based on personalized menu plans
  Arms: Nutritional concept without individual nutritional counselling

SUMMARY:
The PrevA study is designed to evaluate our developed nutritional concept to implement a heart healthy diet. The nutritional concept based on nutrient-optimized daily menu plans for each study day. The plans are personalized according to participants age, gender, and level of physical activity. The PrevA study consists of four periods differing in the energy intake specified by the menu plans.

The study is carried out in a 4-armed parallel design. In group 1, the participants receive the individualized daily plans via the app coupled with the smartwatch to record participants physical activity and heart rate. Groups 2 and 3 receive a printed version of the daily plans with or without personal nutritional advice. The fourth group serves as a control group, which receives general nutritional recommendations but no daily menu plans. During this time, blood samples and urine are collected every four weeks to analyze the study parameters.

DETAILED DESCRIPTION:
Smartphone-based communication technologies are developing rapidly, and the number of so-called mobile health applications is rising. The number of validated and scientifically tested offers is comparatively small. To address this weak point, we developed a personalized nutritional concept to implement a heart-healthy diet. In cooperation with the Preventicus GmbH, Jena, the concept was integrated in an App-based tool. In addition, the app relates to a smartwatch to encourage and track physical activity. The PrevA study will be conducted to evaluate the overall concept.

The nutritional concept based on nutrient-optimized daily menu plans for each study day. The plans are personalized according to participants age, gender, and level of physical activity.

The study is carried out in a 4-armed parallel design. In group 1, the participants receive the individualized daily plans via the app coupled with the smartwatch to record participants physical activity and heart rate. Groups 2 and 3 receive a printed version of the daily plans with or without personal nutritional advice. The fourth group serves as a control group, which receives general nutritional recommendations but no daily menu plans.

In groups 1 to 3, the daily plans are issued in 4 energy levels. At the beginning, the test subjects receive daily plans according to the recommendations for energy intake of the German Nutrition Society (DGE), adapted to their age, gender, and activity level (level 1). After four study weeks, the energy content of the plans is reduced to 85% of the energy intake recommended by the DGE (level 2) and after further four weeks of the PrevA study the energy level is reduced to 70% of the energy intake recommended by the DGE (level 3). Level 4 serves as a stabilization phase and provides the energy content of level 1. The study period extends over a total of 16 study weeks. During this time, blood samples and urine are collected every four weeks to analyze the study parameters. In addition, anthropometric data, data on personal health status and cardiovascular risk profile are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation with documented informed consent
* Willingness and ability to adhere to the study protocol
* Males / female) aged ≥ 20 years and ≤ 51 years
* BMI: ≥ 25 ≤ 35 kg / m2 (obesity grade 1)
* Owning a smartphone (android)
* no or moderate alcohol consumption (≤ 2 glasses / week)
* non-smoker (if possible)

Exclusion Criteria:

Comorbidities:

* Hypercholesterolemia (genetic defect / familial predisposition)
* Diabetes mellitus type 1 or 2
* Thyroid dysfunction (hyper- or hypothyroidism)
* Food intolerance / allergies to ingredients in the study foods
* Medications: lipid-lowering drugs, glucocorticoids
* Dietary supplements: especially n-3 fatty acids, vitamin E.
* Extremely high physical activity (daily)
* Alcohol abuse (daily)
* (smoker) [if there are not enough test persons available, > 7 smokers should be included so that a statistical analysis is possible]
* Uncontrolled organic diseases
* Alcohol, drug or drug abuse
* Participation in other clinical observational studies during or 4 weeks. before starting this study
* Serious behavioral problems, emotional problems or psychiatric problems which the investigator believes would lead to a lack of compliance
* Pregnancy, breastfeeding and unsafe contraception
* Other reasons that are considered important by the investigator

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Body weight | change from baseline after 4, 8, 12, 16 weeks
  Body weight (kg)

SECONDARY OUTCOMES:
Body fat | change from baseline after 4, 8, 12, 16 weeks
  Body fat (%)
Systolic blood pressure | change from baseline after 4, 8, 12, 16 weeks
  systolic pressure (mm Hg)
Diastolic blood pressure | change from baseline after 4, 8, 12, 16 weeks
  diastolic blood pressure (mm Hg)
Basal metabolic rate | change from baseline after 4, 8, 12, 16 weeks
  Basal metabolic rate (kcal per day) - measurement: indirect calorimetry
Total cholesterol (plasma) | change from baseline after 4, 8, 12, 16 weeks
  Total cholesterol (mmol/l)
LDL cholesterol (plasma) | change from baseline after 4, 8, 12, 16 weeks
  LDL cholesterol (mmol/l)
HDL cholesterol (plasma) | change from baseline after 4, 8, 12, 16 weeks
  HDL cholesterol (mmol/l)
Triacylglycerides (plasma) | change from baseline after 4, 8, 12, 16 weeks
  Triacylglycerides (mmol/l)
Glucose (fasting) (serum) | change from baseline after 4, 8, 12, 16 weeks
  Glucose (mmol/l)
Insulin (fasting) (serum) | change from baseline after 4, 8, 12, 16 weeks
  Insulin (mU/l)
HbA1c (serum) | change from baseline after 4, 8, 12, 16 weeks
  HbA1c (%)
alpha prothrombin time (serum) | change from baseline after 4, 8, 12, 16 weeks
  alpha prothrombin time (s)
Fibrinogen (serum) | change from baseline after 4, 8, 12, 16 weeks
  Fibrinogen (g/l)
High sensitive c-reactive protein (plasma) | change from baseline after 4, 8, 12, 16 weeks
  High sensitive c-reactive protein (mg/l)
Homocysteine (serum) | change from baseline after 4, 8, 12, 16 weeks
  Homocysteine (µmol/l)
Triiodothyronine (plasma) | change from baseline after 16 weeks
  Triiodothyronine fT3 (pmol/l)
Thyroxine (plasma) | change from baseline after 16 weeks
  Thyroxine fT4 (pmol/l)
Thyroid-stimulating hormone (plasma) | change from baseline after 16 weeks
  Thyroid-stimulating hormone (mU/l)
Parathyroid hormone (plasma) | change from baseline after 16 weeks
  Parathyroid hormone (ng/l)
Alkaline phosphatase (serum) | change from baseline after 16 weeks
  Alkaline phosphatase (µg/l)
Osteocalcin (serum) | change from baseline after 16 weeks
  Osteocalcin (ng/ml)
Uric acid (plasma) | change from baseline after 16 weeks
  Uric acid (µmol/l)
Alanine aminotransferase (plasma) | change from baseline after 4, 8, 12, 16 weeks
  Alanine aminotransferase (µmol/l*s)
Aspartate transaminase (plasma) | change from baseline after 4, 8, 12, 16 weeks
  Aspartate transaminase (µmol/l*s)
Cholinesterase (plasma) | change from baseline after 4, 8, 12, 16 weeks
  Cholinesterase (µmol/l*s)
Gamma-glutamyltransferase (plasma) | change from baseline after 4, 8, 12, 16 weeks
  Gamma-glutamyltransferase (µmol/l*s)
Lactate dehydrogenase (plasma) | change from baseline after 4, 8, 12, 16 weeks
  Lactate dehydrogenase (µmol/l*s)
Fatty acid distribution in plasma lipids (plasma) | change from baseline after 4, 8, 12, 16 weeks
  Fatty acid distribution in plasma lipids (% fatty acid methyl esters)
Fatty acid distribution in erythrocyte lipids (erythrocytes) | change from baseline after 4, 8, 12, 16 weeks
  Fatty acid distribution in erythrocyte lipids (% fatty acid methyl esters)
Vitamin A (serum) | change from baseline after 16 weeks
  Vitamin A (mmol/l)
Vitamin D (plasma) | change from baseline after 16 weeks
  Vitamin D (nmol/l)
Vitamin E (serum) | change from baseline after 16 weeks
  Vitamin E (µmol/l)
Vitamin B1 (serum) | change from baseline after 16 weeks
  Vitamin B1 (nmol/l)
Vitamin B2 (serum) | change from baseline after 16 weeks
  Vitamin B2 (nmol/l)
Vitamin B6 (serum) | change from baseline after 16 weeks
  Vitamin B6 (nmol/l)
Vitamin B12 (plasma) | change from baseline after 16 weeks
  Vitamin B12 (pmol/l)
Holo-transcobalamin (plasma) | change from baseline after 16 weeks
  Holo-transcobalamin (pmol/l)
Folic acid (plasma) | change from baseline after 16 weeks
  Folic acid (µg/l)
Vitamin H (serum) | change from baseline after 16 weeks
  Vitamin H (ng/l)
Vitamin C (plasma) | change from baseline after 16 weeks
  Vitamin C (mg/l)
Calcium (plasma) | change from baseline after 16 weeks
  Calcium (mmol/l)
Potassium (plasma) | change from baseline after 16 weeks
  Potassium (mmol/l)
Iron (plasma) | change from baseline after 4, 8, 12, 16 weeks
  Iron (µmol/l)
Ferritin (plasma) | change from baseline after 4, 8, 12, 16 weeks
  Ferritin (µg/l)
Transferrin (plasma) | change from baseline after 4, 8, 12, 16 weeks
  Transferrin (g/l)
Iodine (serum) | change from baseline after 16 weeks
  Iodine (µmol/l)
Selenium (serum) | change from baseline after 16 weeks
  Selenium (µmol/l)
Zinc (serum) | change from baseline after 16 weeks
  Zinc (µmol/l)

OTHER OUTCOMES:
Creatinine (24 h urine) | change from baseline after 16 weeks
  Creatinine (mmol/l)
Albumine (24 h urine) | change from baseline after 16 weeks
  Albumine (mg/l)
Selenium (24 h urine) | change from baseline after 16 weeks
  Selenium (µmol/24 h)
Zinc (24 h urine) | change from baseline after 16 weeks
  Zinc (µmol/24 h)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Dawczynski, PhD, Principal Investigator — Friedrich-Schiller-University
Locations (1):
- Friedrich-Schiller University, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No